CLINICAL TRIAL: NCT06726863
Title: A Phase 1, Randomized, Open-label Study to Characterize the Pharmacokinetics, Pharmacodynamics, and Safety of Vamifeport After Multiple Oral Administration of One Immediate-release Formulation and After Single and Multiple Oral Administration of Two Prolonged-release Formulations in Healthy Adult Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics of Two Prolonged-release Formulations of Vamifeport in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CSL624_1005
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Oral ferroportin inhibitor; Ferroportin transporter; Iron overload; Iron metabolism
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Intervention Model Description: This is a 4-treatment period study that uses three different models: Treatment Period 1 will be a single-arm model, Treatment Period 2 will be a parallel-group model, and Treatment Periods 3 and 4 will be crossover models.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Treatment Period 1: Vamifeport IR Formulation Dose Level 1 (Experimental): Participants will receive multiple doses of Vamifeport Immediate-release (IR) formulation at Dose level 1.
  Interventions: Drug: Vamifeport IRF
- Treatment Period 2: Vamifeport PR1 Dose Level 2 (Experimental): Participants will receive multiple doses of Vamifeport Prolonged-release formulation 1 (PR1) at Dose level 2.
  Interventions: Drug: Vamifeport PR1
- Treatment Period 2: Vamifeport PR2 Dose Level 2 (Experimental): Participants will receive multiple doses of Vamifeport Prolonged-release formulation 2 (PR2) at Dose level 2.
  Interventions: Drug: Vamifeport PR2
- Treatment Period 3: Vamifeport PR1 Dose Level 3 (Experimental): Participants will receive a single dose of Vamifeport PR1 at Dose level 3.
  Interventions: Drug: Vamifeport PR1
- Treatment Period 3: Vamifeport PR2 Dose Level 3 (Experimental): Participants will receive a single dose of Vamifeport PR2 at Dose level 3.
  Interventions: Drug: Vamifeport PR2
- Treatment Period 4: Vamifeport PR1 Dose Level 3 (Experimental): Participants will receive a single dose of Vamifeport PR1 at Dose level 3.
  Interventions: Drug: Vamifeport PR1
- Treatment Period 4: Vamifeport PR2 Dose Level 3 (Experimental): Participants will receive a single dose of Vamifeport PR2 at Dose level 3.
  Interventions: Drug: Vamifeport PR2

INTERVENTIONS:
Drug: Vamifeport IRF — Vamifeport IRF will be administered orally as per the dosing levels and formulations for respective treatment periods.
  Other Names: CSL624
  Arms: Treatment Period 1: Vamifeport IR Formulation Dose Level 1
Drug: Vamifeport PR1 — Vamifeport PR1 will be administered orally as per the dosing levels and formulations for respective treatment periods.
  Other Names: CSL624
  Arms: Treatment Period 2: Vamifeport PR1 Dose Level 2; Treatment Period 3: Vamifeport PR1 Dose Level 3; Treatment Period 4: Vamifeport PR1 Dose Level 3
Drug: Vamifeport PR2 — Vamifeport PR2 will be administered orally as per the dosing levels and formulations for respective treatment periods.
  Other Names: CSL624
  Arms: Treatment Period 2: Vamifeport PR2 Dose Level 2; Treatment Period 3: Vamifeport PR2 Dose Level 3; Treatment Period 4: Vamifeport PR2 Dose Level 3

SUMMARY:
This is a phase 1, single-center, randomized, open-label study to characterize the pharmacokinetics (PK), pharmacodynamics (PD), and safety of vamifeport after multiple oral administrations of one immediate-release (IR) formulation and after single and multiple oral administrations of two prolonged-release (PR) formulation in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to (>=) 18 to less than or equal to (<=) 60 years when providing written informed consent.
* Healthy, as determined by the investigator based on review of defined assessments during Screening.
* Body weight between 50 and 100 kilograms (kg) (inclusive) and body mass index within the range 18.0 to 32.0 kg per meter squared (kg/m2) (inclusive) at Screening and Day -1.

Exclusion Criteria:

* Any clinically relevant abnormal 12-lead ECG finding at Screening or Day -1 (as deemed by the investigator).
* Serum ferritin of < 30 nanograms per milliliter (ng/mL) or > 300 ng/mL for assigned male at birth (AMAB) subjects or <16 ng/mL or > 300 ng/mL for assigned female at birth (AFAB) subjects at Screening or Day -1.
* Hemoglobin < 13 grams per deciliter (g/dL) (8.1 millimoles per liter [mmol/L]) for AMAB subjects or 12 g/dL (7.5 mmol/L) for AFAB subjects at Screening or Day -1.
* Blood draw or donation of blood (>= 450 mL) within 3 months before Screening, plasma from 2 weeks before Screening, or platelets from 6 weeks before Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration-time course profiles of vamifeport | Treatment Period (TP) 2: Before and after dosing on Day 4 (up to 12 hours), Day 8 (up to 48 hours), Before dosing on Day 5, 6, 7 TP 3: Before and after dosing on Day 13 (up to 48 hours) TP 4: Before and after dosing on Day 16 (up to 48 hours)
Maximum plasma concentration (Cmax) of first and last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP2: Before, and up to 48 hours after, both the first and the last dose
Time to reach Cmax (Tmax) of first and last dose vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after, both the first and the last dose
Area under the plasma concentration curve from time zero to 12 hours (AUC0-12) of first and last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after, both the first and the last dose
Trough concentration (Ctrough) of first dose of vamifeport PR1 and PR2 in Treatment Period 2 | Before and up to 24 hours after the first dose in TP2
AUC from time zero to infinity (AUC0-inf) of last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after last dose
AUC from time zero to time tlast (AUC0-last) of last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after last dose
AUC from time zero to 8 hours (AUC0-8) and 24 hours (AUC0-24) of last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 8 and 24 hours after last dose
Plasma concentration at 12 hours (Conc [t=12]) of last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before and up to 12 hours after last dose
Apparent clearance (CL/F) of last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after last dose
Apparent volume of distribution at steady state (Vss/F) of last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after last dose
Accumulation ratio (Rac) of Cmax between first and last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after first and last dose
Rac(Ctrough/Conc[t=12]) between first and last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 12 hours after first and last dose
Rac (AUC0-12) between first and last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 12 hours after first and last dose
Half-life (t1/2) after last dose of vamifeport PR1 and PR2 in Treatment Period 2 | TP 2: Before, and up to 48 hours after last dose
Cmax of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
Tmax of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
AUC0-inf of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
AUC0-last of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
AUC0-8, AUC0-12 and AUC0-24 of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 8, 12 and 24 hours after dosing, in TP3 and TP4
Plasma Concentration at 8 hours (Conc [t=8]), 12 hours (Conc [t=12]) and 24 hours (Conc [t=24]) of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 8, 12 and 24 hours after dosing, in TP3 and TP4
CL/F of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
t1/2 of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
Apparent volume of distribution (Vz/F) of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4

SECONDARY OUTCOMES:
Number of participants with treatment-emergent (TE): adverse event (AE), AE by severity, AE related to vamifeport, and serious AE | Up to 25 days after treatment
Percentage of participants with TEAE, AE by severity, AE related to vamifeport, and serious AE | Up to 25 days after treatment
Number of participants with clinically significant change from Baseline in clinical laboratory safety tests, 12 lead Electrocardiogram (ECG), and vital signs | At baseline and up to 25 days after treatment
  The clinical laboratory safety tests include biochemistry, hematology, urinalysis.
AUC0-24 of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 24 hours after dosing, in TP3 and TP4
  Comparison of AUC0-24 between PR1 and PR2
AUC0-12 of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 12 hours after dosing, in TP3 and TP4
  Comparison of AUC0-12 between PR1 and PR2
AUC0-inf of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
  Comparison of AUC0-inf between PR1 and PR2
Conc (t=12) of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 12 hours after dosing, in TP3 and TP4
  Comparison of conc(t=12) between PR1 and PR2
Conc (t=24) of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 24 hours after dosing, in TP3 and TP4
  Comparison of conc(t=24) between PR1 and PR2
Cmax of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
  Comparison of cmax between PR1 and PR2
Tmax of vamifeport PR1 and PR2 in Treatment Period 3 and 4 | Before and up to 48 hours after dosing, in TP3 and TP4
  Comparison of tmax between PR1 and PR2
Absolute values of serum iron | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Absolute values of transferrin saturation (TSAT) | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Change from baseline of serum iron | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Change from baseline of TSAT | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Maximum percentage change from baseline (Emax) of serum iron | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Emax of TSAT | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Time to Emax (TEmax) of serum iron | Before and up to 48 hours after dosing in TP2, TP3 and TP4
TEmax of TSAT | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Time below baseline of serum iron | Before and up to 48 hours after dosing in TP2, TP3 and TP4
Time below baseline of TSAT | Before and up to 48 hours after dosing in TP2, TP3 and TP4
AUC below baseline of serum iron | Before and up to 48 hours after dosing in TP2, TP3 and TP4
AUC below baseline of TSAT | Before and up to 48 hours after dosing in TP2, TP3 and TP4

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Investigator Site 82600083, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.